CLINICAL TRIAL: NCT06378463
Title: Improving Outcome Through Improving Cognition in Severe Mental Illness: Cognitive Remediation Training Combined With Transcranial Direct Current Stimulation, a Randomized, Sham-controlled, Multi-center Trial
Brief Title: Cognitive Remediation and Transcranial Direct Current Stimulation in Severe Mental Illness (SMI)
Acronym: HEADDSET+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Groningen (Other)
Collaborators: Stichting Cosis (Unknown); Lentis Psychiatric Institute (Other); GGZ Friesland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSY-2324-S-0362
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Severe Mental Illness
Keywords: Cognitive training; Cognitive functioning; Cognitive rehabilitation; Cognitive remediation; Functional recovery; Community recovery; Non-invasive brain stimulation; transcranial Electrical Stimulation; transcranial Direct Current Stimulation
MeSH Terms: conditions — Mental Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Intervention Model Description: This is a pragmatic triple-blinded, randomized, sham-controlled trial, following a non-concurrent multiple baseline design, with the participants serving as their own control. Participants will be randomized over two groups: CIRCuiTS +sham tDCS (group 1), or CIRCuiTS + active tDCS (group 2). The trial will start with a first measurement (T0), followed by a waiting period of 16 weeks and a second measurement (T1). The waiting period serves as the control condition (service users are their own control). Next, the participants will be allocated to 16-20 weeks of either CIRCuiTS + sham tDCS or CIRCuiTS + active tDCS. This period of 16-20 weeks is not fixed as it depends upon how fast participants go through the program. This is followed by a third measurement after treatment (T2). There will be a fourth measurement six months after the end of the intervention (T3).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomly assigned to CR + sham tDCS (group 1) or CR + active tDCS (group 2) with a 1:1 allocation as per a computer-generated randomization plan using permuted blocks of random sizes. The block sizes will not be disclosed to ensure concealment. As such, both the researcher as the participant can stay blind to the tDCS treatment condition. Also, the assessors who will do neuropsychological tests are blind to the condition the participant is in and are blind to the type and aim of the treatment. After finishing measurement T2, the participants can indicate if they suspect to have experienced either the real or the sham tDCS treatment. The patients will be informed about the type of treatment they have received when all participants completed measurement T3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active tDCS + CR (Active Comparator): For active tDCS, the current will be 2 mA and will be administered for 20 min with a fade-in/out of 30 s. The anode will be positioned at Fp1 and the cathode at C3, following the 10-20 system.
  Interventions: Other: Cognitive remediation + active tDCS
- sham tDCS + CR (Sham Comparator): For the sham tDCS, the fade-in will be identical as for the active tDCS. After 30 s the current will fade-out over 30 s. In addition to those above, a standard control pulse, with no therapeutic effect, will be frequently sent to monitor electric conductivity (~ 0.02mA in duration of 3 s, send every 0.55 s). The anode will be positioned at Fp1 and the cathode at C3, following the 10-20 system.
  Interventions: Other: Cognitive remediation + sham tDCS

INTERVENTIONS:
Other: Cognitive remediation + active tDCS — The cognitive remediation program "Computerised Interactive Remediation of Cognition - a Training for Schizophrenia" (CIRCuiTS) improves cognitive and metacognitive skills and strategies and is specifically aimed at the generalization of newly learnt skills to daily life. This method also offers the possibility to personalize the training program based on individual goals and cognitive functioning of the service user.
  Transcranial Direct Current Stimulation is used to promote neural plasticity, which applies a small electrical current over the cortex. This can alter the excitability of neurons, such that it increases or decreases spontaneous network activity. When applied to fronto-parietal neural networks simultaneously with their engagement in cognitive tasks of CIRCuiTS, it is expected that plasticity of these networks will be modulated, resulting in improvements in cognitive functioning.
  In this condition, participants will receive active brain stimulation.
  Arms: active tDCS + CR
Other: Cognitive remediation + sham tDCS — The cognitive remediation program "Computerised Interactive Remediation of Cognition - a Training for Schizophrenia" (CIRCuiTS) improves cognitive and metacognitive skills and strategies and is specifically aimed at the generalization of newly learnt skills to daily life. This method also offers the possibility to personalize the training program based on individual goals and cognitive functioning of the service user.
  Transcranial Direct Current Stimulation is used to promote neural plasticity, which applies a small electrical current over the cortex. This can alter the excitability of neurons, such that it increases or decreases spontaneous network activity. When applied to fronto-parietal neural networks simultaneously with their engagement in cognitive tasks of CIRCuiTS, it is expected that plasticity of these networks will be modulated, resulting in improvements in cognitive functioning.
  In this condition, participants will receive sham brain stimulation.
  Arms: sham tDCS + CR

SUMMARY:
Seven per cent of patients suffering from severe mental illness (SMI) need long-term intensive treatment and support in a clinical setting or sheltered living. These service users often experience problems on multiple domains, such as persistent complaints as a result of medication resistance, physical health problems and self-care, psychosocial and cognitive dysfunctioning. Cognitive remediation (CR) training is a type of training aimed at improving thinking abilities (cognitive functioning) and daily functioning. However, we don't yet know if CR training can also help people with SMI who need supported housing due to their severe cognitive and daily living problems. In this project, we are investigating whether we can improve daily functioning in this group by using a form of CR training that focuses on learning new cognitive skills and how to use these new skills in everyday life. Additionally, we are exploring whether combining CR training with mild brain stimulation (transcranial Direct Current Stimulation) can enhance the effects of CR training.

DETAILED DESCRIPTION:
A fundamental challenge for many people with severe mental illness (SMI) is dealing with the impact of cognitive impairments in daily life functioning. A possible treatment approach is cognitive remediation training (CR), a training developed to target cognitive deficits with the ultimate aim to improve daily functioning. Participants engage in cognitive exercises, learn more about their own cognition and the use of (cognitive) strategies to compensate for deficits. However, in people with SMI, abnormal synaptic plasticity is observed. This might hinder newly learned cognitive skills to sustain and limit the benefits from CR. For this reason, people with SMI may benefit from the combination of CR with a method that may promote neural plasticity: transcranial direct current stimulation (tDCS).

In a pragmatic, triple-blinded, randomized, sham-controlled, multi-center trial with a multiple baseline design, we will investigate the effectiveness of combining CR and tDCS in helping participants reach personal goals, minimizing problems in daily functioning and improving cognitive functioning. 126 service users with SMI will receive 16-20 weeks of twice-weekly CR combined with active (N=63) or sham tDCS (N=63). We will perform functional, cognitive, and clinical outcome assessments at baseline, after a 16-week waiting period, post-treatment and 6-months post-treatment and compare the effects within-participants (waiting period vs. treatment period) and between-participants (CR+active tDCS vs. CR+sham tDCS). Further, an optional in-depth interview will be conducted post-intervention (T2) to investigate subjective experiences of CR and its perceived effect on metacognition, daily functioning, helpful components, and areas for improvement.

This multi-center trial will evaluate whether CR on its own and whether CR in combination with tDCS can be a clinically relevant addition to further enhance recovery through enhancing service users' goal attainment, daily functioning and cognitive performance. In case results of this trial confirm our hypotheses, it may be recommended to include the combined information in the guidelines for SMI care and to implement the method in standardized care.

ELIGIBILITY:
Inclusion Criteria:

* A psychiatric disorder that requires care/treatment (no remission of positive, negative and cognitive symptoms);
* Severe disabilities in social and/or societal functioning (no functional remission);
* Disabilities are the result of a psychiatric disorder;
* Disabilities are structural (at least several years);
* Coordinated professional care is necessary to realize a treatment plan;
* Adults between the age of 18 and 65;
* Sufficient written and oral mastery of the Dutch language.

Exclusion Criteria:

* Having previously received CIRCuiTS;
* Metal implants inside the skull or eye;
* Severe scalp skin lesions;
* A history of previous seizures;
* Alcohol or drug abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Independent Living Skills Survey self- and observer-rated questionnaire (ILSS) | Baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment
  The Independent Living Skills Survey (ILSS) is a questionnaire that measures the basic functional living skills of individuals with SMI. The ILSS will be completed by the participant and by the participant's case manager.
Goal Attainment Scale (GAS) | Baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment
  This questionnaire is a measure to capture self-reported recovery goals in a structured way, which has also been used in rehabilitation practice. Based upon an interview, the participant defines up to three personal recovery goals that can be scored and weighted on importance and difficulty for which a scoring manual is available.
Social Functioning Scale (SFS) | Baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment
  The SFS is a standard measure that was developed and validated for people with schizophrenia and includes the following subscales: social engagement or withdrawal, interpersonal functioning, current social activities, recreational activities, independence-competence, independence-performance, and employment.
Behapp application | Throughout the entire study period, up to 16 months (including baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment)
  Behapp is a smartphone app that was developed to objectively and passively measure sociability and social exploration. After installation, Behapp will continuously monitor measures of communication events (e.g., incoming and outgoing phone calls), app activity (e.g., social media or entertainment apps), and location via GPS. Data are encrypted before saving on the participants' device and deleted immediately after uploading to the secured data server. The content of calls, SMS messages, and apps will not be registered, collected, or saved by Behapp.

SECONDARY OUTCOMES:
Controlled Oral World Association Task (COWAT) | Baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment
  The COWAT is a test for verbal fluency and speed of processing. Participants have to name as many words as possible within a time span of 60 seconds, beginning with a given letter.
Trail Making Test (TMT) | Baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment
  The Trail Making Test assesses visual search abilities, processing speed, and mental flexibility. Participants are provided with a sheet of paper, containing only digits or digits and letters, and are instructed to connect them in increasing order.
Digit span (forward & backward) | Baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment
  The Digit Span forward is a test for immediate auditory attention. The Digit Span backward is a test for working memory. The test leader reads sequences of digits out loud, gradually increasing the digit span. The participant is asked to repeat the digits in the same order (forward) or reverse order (backward).
Wechsler Memory Scale - Visual Reproduction I and II | Baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment
  The Visual Reproduction subtest of the Wechsler Memory Scale (WMS) assesses visual memory for abstract designs. During this task, participants are presented with a series of designs. Each design is displayed for 10 seconds, after which the participant is asked to reproduce it from memory. After 30 minutes, a recognition task of the same designs is administered.
Stroop Color and Word Task (SCWT) | Baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment
  The SCWT is used to test speed of processing, cognitive flexibility, and cognitive control. The participants first perform a basic task, which is reading names of colors. The performance on this task is compared with the performance on a task in which the ink color of incongruent color words has to be named. Hence, a habitual response needs to be suppressed in support of an unusual one. The increase in time taken to perform the latter task compared with the basic task is referred to as "the Stroop interference effect" and provides a general measure of executive functioning.
15 Word Test (15-WT) | Baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment
  The 15-WT learning task is a test for verbal memory. The test leader reads 15 words out loud and participants are asked to recall as many words as possible. This procedure is repeated for four times.
Behavioral Assessment of the Dysexecutive System (BADS) - Key Search task | Baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment
  The Key search task is a subtest of the BADS, a test battery used to evaluate executive functions. In this task, participants are asked to plan a search route for an imaginary lost key within a field.
Cognitive Failure Questionnaire (CFQ) | Baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment
  The CFQ is a questionnaire to measure subjective cognitive functioning. The scale includes 25 questions that represent the cognitive subdomains attention and memory.
Self-Evaluation of Negative Symptoms (SNS) | Baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment
  The SNS questionnaire assesses negative symptoms from the perspective of the service user.
DEX self/informant | Baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment
  The DEX questionnaire is a 20-item measure used to evaluate subjective cognitive performance, focusing on problems related to planning and organization. There are two versions of the questionnaire: one to be completed by the participant and the other by their case manager.
General Self-Efficacy Scale (GSES) | Baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment
  The GSES is a measure used to assess self-efficacy, the degree to which the respondent perceives himself or herself as capable of attaining goals, overcoming challenges, and performing well on tasks.
Nurses' Observation Scale of Cognitive Abilities (NOSCA) | Baseline (16 weeks before start of treatment), pre-treatment, post-treatment (after 16-20 weeks of treatment) and 6-months post-treatment
  The NOSCA is a behavioral rating scale to examine cognitive abilities in service users. The scale comprises eight subscales, representing subdomains of cognition. The answers are based on observations of a participants' case manager.
In-depth interview | Post-treatment (after 16-20 weeks of treatment)
  The in-depth interview aims to understand service users' metacognitive skills and subjective experiences. An adapted version of the Metacognition Assessment Scale (MAS-A) is used. Higher scores on each subscale (self-reflectivity, understanding the other's mind, decentration, and mastery) indicate a greater ability to form complex representations of oneself and others. The MAS-A is used to score the answers on the Indiana Psychiatric Illness Interview (IPII), a semi-structured interview designed to examine spontaneous metacognitive thoughts that lasts 30 to 60 minutes. We revised the IPII to emphasize cognitive experiences over illness experiences and to evaluate metacognitive ability.

CONTACTS AND LOCATIONS:
Overall Officials: Lisette van der Meer, PhD, Principal Investigator — Department of Clinical and Developmental Neuropsychology
Locations (3):
- Netherlands (3):
  - Cosis, Assen, Drenthe
  - Lentis, Zuidlaren, Drenthe
  - GGZ Friesland, Leeuwarden, Provincie Friesland

IPD SHARING:
Plan to Share IPD: No